CLINICAL TRIAL: NCT04370782
Title: A Randomized Study Evaluating the Safety and Efficacy of Hydroxychloroquine and Zinc in Combination With Either Azithromycin or Doxycycline for the Treatment of COVID-19 in the Outpatient Setting
Brief Title: Hydroxychloroquine and Zinc With Either Azithromycin or Doxycycline for Treatment of COVID-19 in Outpatient Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Francis Hospital, New York (Other)
Responsible Party: Principal Investigator, Avni Thakore MD, Principal Investigator, St. Francis Hospital, New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-21
Record Dates: First submitted 2020-04-26; First posted 2020-05-01 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
Keywords: coronavirus; hydroxychloroquine; zinc sulfate
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Hydroxychloroquine; Azithromycin; Zinc Sulfate; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm 1 (Experimental): Hydroxychloroquine
  Azithromycin
  Zinc sulfate
  Interventions: Drug: Hydroxychloroquine; Drug: Azithromycin; Drug: Zinc Sulfate
- Experimental Arm 2 (Experimental): Hydroxychloroquine
  Doxycycline
  Zinc sulfate
  Interventions: Drug: Hydroxychloroquine; Drug: Zinc Sulfate; Drug: Doxycycline

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 400mg twice a day (BID) on day 1, followed by 200mg BID for days 2-5
Drug: Azithromycin — Azithromycin 500mg on day 1, followed by 250mg once daily for days 2-5
  Arms: Experimental Arm 1
Drug: Zinc Sulfate — Zinc sulfate 220mg once daily for 5 days
Drug: Doxycycline — Doxycycline 200 mg once daily for 5 days
  Arms: Experimental Arm 2

SUMMARY:
This is a randomized, open-label trial to assess the safety and efficacy of hydroxychloroquine, and zinc in combination with either azithromycin or doxycycline in a higher risk COVID-19 positive outpatient population.

DETAILED DESCRIPTION:
COVID-19 is an aggressive and contagious virus, found to have high mortality especially in persons with comorbidities (Age>60, hypertension [HTN], diabetes mellitus [DM], Cancer, and otherwise immunocompromised). Zinc is a supplement with possible antiviral properties, having been shown to have effect in the common cold, many of which are due to coronavirus. In addition, elderly patients and patients with co-morbidities have high incidence of zinc deficiency. We are repleting zinc in all patients and studying its direct effect in combination with hydroxychloroquine, and an antibiotic, either azithromycin or doxycycline to see if there is enhanced treatment efficacy in early COVID-19 infection and assess the safety of these two regimen.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand informed consent.
* High initial clinical suspicion by physician based on signs and symptoms (fever, cough, myalgias, fatigue, shortness of breath) followed by RT-PCR for confirmation of COVID-19 diagnosis
* Any gender
* Age 60 years and older
* Age 30-59 years with one or more of the following:

  * abnormal lung exam
  * abnormal oxygen staturation <95%
  * abnormal chest x-ray or chest CT
  * persistent fever >100.4 degrees Fahrenheit upon arrival to Emergency department (ED)
  * one of the following co-morbidities: hypertension, diabetes mellitus, history of coronary artery disease, chronic kidney disease (CKD), asthma, chronic obstructive pulmonary disease, current or former smoker, or morbid obesity (Body Mass Index ≥35)

Exclusion Criteria:

* Pregnant or breastfeeding female
* Severe COVID-19 requiring admission for inpatient treatment
* Need for any oxygen supplementation
* Need for mechanical ventilatory support
* History of oxygen supplementation dependency
* History of cancer with ongoing chemotherapy or radiation therapy
* Concurrent antimicrobial therapy
* Known hypersensitivity to hydroxychloroquine or other 4-aminoquinoline compounds
* Already taking hydroxychloroquine or chloroquine within 1 month
* Known G6-PD deficiency
* History of retinopathy
* History of current cardiac diseases (heart failure, ventricular arrhythmias, Left bundle branch block and/or Right bundle branch block, QTc prolongation >480ms), or family history of sudden cardiac death
* Ongoing use of drugs that prolong the QTc interval (antipsychotics, antidepressants, class I and III antiarrhythmics, triptans)
* Severe renal disease: glomerular filtration rate (GFR) <30ml/min
* Severe hepatic impairment (elevated total bilirubin >2 mg/dL, decreased albumin <2.8 g/dL, signs of jaundice and ascites.)
* Active alcohol abuse (>5 drinks per day or >20 drinks per week.)
* Seizure disorder, currently on medications
* Known hypersensitivity to any tetracyclines.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Time to Resolution of Symptoms relative to baseline (day 1 of trial) | Day 5
  Patients will be assessed on day 5 for when COVID-19 symptoms completely resolve compared to baseline (day 1 of trial)
Time to Resolution of Symptoms relative to baseline (day 1 of trial) | Day 14
  Patients will be assessed on day 14 for when COVID-19 symptoms completely resolve compared to baseline (day 1 of trial)
Time to Resolution of Symptoms relative to baseline (day 1 of trial) | Day 21
  Patients will be assessed on day 21 for when COVID-19 symptoms completely resolve compared to baseline (day 1 of trial)
Number of participants hospitalized and/or requiring repeat ER visits | 21 days
  Number of participants hospitalized and/or requiring repeat ER visits related to COVID-19 complications
ICU Length of Stay | Until Discharged up to 30 days
  If hospitalized, number of participants admitted to the ICU, and number of days in the ICU
Ventilator | Until extubated up to 30 days
  If placed on ventilator, number of days on a ventilator

SECONDARY OUTCOMES:
Severity of symptoms | Day 5, Day 14, and Day 21
  Severity of symptoms evaluated at day 5, day 14, and day 21 scored by the participant for feverishness, sore throat, cough, shortness of breath, myalgias. (0 =none; 1 = mild; 2 = moderate; 3 = severe)
Number of participants with adverse events due to drug regimen | 21 days
  Number of participants with adverse events due to drug regimen
Number of participants with QTc prolongation >500ms | Days 1 thru 5, Day 10, Day 21
  Assess all patients to evaluate for QTc prolongation >500ms

CONTACTS AND LOCATIONS:
Overall Officials: Avni Thakore, MD, Principal Investigator — Saint Francis Hospital
Locations (1):
- St Francis Hospital, Roslyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Background] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Background] Devaux CA, Rolain JM, Colson P, Raoult D. New insights on the antiviral effects of chloroquine against coronavirus: what to expect for COVID-19? Int J Antimicrob Agents. 2020 May;55(5):105938. doi: 10.1016/j.ijantimicag.2020.105938. Epub 2020 Mar 12. PMID 32171740
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Kim AHJ, Sparks JA, Liew JW, Putman MS, Berenbaum F, Duarte-Garcia A, Graef ER, Korsten P, Sattui SE, Sirotich E, Ugarte-Gil MF, Webb K, Grainger R; COVID-19 Global Rheumatology Alliance. A Rush to Judgment? Rapid Reporting and Dissemination of Results and Its Consequences Regarding the Use of Hydroxychloroquine for COVID-19. Ann Intern Med. 2020 Jun 16;172(12):819-821. doi: 10.7326/M20-1223. Epub 2020 Mar 30. Erratum In: Ann Intern Med. 2020 Jun 16;172(12):844. doi: 10.7326/L20-0417. PMID 32227189
- [Background] Wu C, Liu Y, Yang Y, Zhang P, Zhong W, Wang Y, Wang Q, Xu Y, Li M, Li X, Zheng M, Chen L, Li H. Analysis of therapeutic targets for SARS-CoV-2 and discovery of potential drugs by computational methods. Acta Pharm Sin B. 2020 May;10(5):766-788. doi: 10.1016/j.apsb.2020.02.008. Epub 2020 Feb 27. PMID 32292689
- [Background] Korant BD, Butterworth BE. Inhibition by zinc of rhinovirus protein cleavage: interaction of zinc with capsid polypeptides. J Virol. 1976 Apr;18(1):298-306. doi: 10.1128/JVI.18.1.298-306.1976. PMID 176466
- [Background] Katz E, Margalith E. Inhibition of vaccinia virus maturation by zinc chloride. Antimicrob Agents Chemother. 1981 Feb;19(2):213-7. doi: 10.1128/AAC.19.2.213. PMID 7347557
- [Background] Kumel G, Schrader S, Zentgraf H, Daus H, Brendel M. The mechanism of the antiherpetic activity of zinc sulphate. J Gen Virol. 1990 Dec;71 ( Pt 12):2989-97. doi: 10.1099/0022-1317-71-12-2989. PMID 2177090
- [Background] Suara RO, Crowe JE Jr. Effect of zinc salts on respiratory syncytial virus replication. Antimicrob Agents Chemother. 2004 Mar;48(3):783-90. doi: 10.1128/AAC.48.3.783-790.2004. PMID 14982765
- [Background] Eby GA, Davis DR, Halcomb WW. Reduction in duration of common colds by zinc gluconate lozenges in a double-blind study. Antimicrob Agents Chemother. 1984 Jan;25(1):20-4. doi: 10.1128/AAC.25.1.20. PMID 6367635
- [Background] te Velthuis AJ, van den Worm SH, Sims AC, Baric RS, Snijder EJ, van Hemert MJ. Zn(2+) inhibits coronavirus and arterivirus RNA polymerase activity in vitro and zinc ionophores block the replication of these viruses in cell culture. PLoS Pathog. 2010 Nov 4;6(11):e1001176. doi: 10.1371/journal.ppat.1001176. PMID 21079686
- [Background] Singh M, Das RR. Zinc for the common cold. Cochrane Database Syst Rev. 2013 Jun 18;(6):CD001364. doi: 10.1002/14651858.CD001364.pub4. PMID 23775705
- [Background] Bao S, Knoell DL. Zinc modulates airway epithelium susceptibility to death receptor-mediated apoptosis. Am J Physiol Lung Cell Mol Physiol. 2006 Mar;290(3):L433-41. doi: 10.1152/ajplung.00341.2005. Epub 2005 Nov 11. PMID 16284213
- [Background] Xue J, Moyer A, Peng B, Wu J, Hannafon BN, Ding WQ. Chloroquine is a zinc ionophore. PLoS One. 2014 Oct 1;9(10):e109180. doi: 10.1371/journal.pone.0109180. eCollection 2014. PMID 25271834